CLINICAL TRIAL: NCT04145063
Title: Ureteric Stenting Versus Non-stenting Following Uncomplicated Ureteroscopic Lithotripsy: A Prospective Randomized Trial
Brief Title: Ureteric Stenting Versus Non-stenting Following Uncomplicated Ureteroscopic Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Saddam Al Demour, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sad2019
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Ureter Stone
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- uncomplicated ureteroscopic lithotripsy with DJ-US (No Intervention): Following uncomplicated uretroscopic lithotripsy, a double J uretric stent will be placed (usually the standard of care)
- uncomplicated ureteroscopic lithotripsy without US (Active Comparator): Following uncomplicated uretroscopic lithotripsy no uretric stent will be placed
  Interventions: Other: no stent
- uncomplicated ureteroscopic lithotripsy with DJ-US-string (No Intervention): Following uncomplicated uretroscopic lithotripsy, a double J uretric stent with an extraxtion string will be placed

INTERVENTIONS:
Other: no stent — following uretroscopy, no stent will be placed
  Arms: uncomplicated ureteroscopic lithotripsy without US

SUMMARY:
This study aims to compare three groups of patients who underwent uncomplicated ureteroscopic lithotripsy (URSL) to evaluate whether stents could be eliminated after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* unilateral ureteric stones managed by ureteroscopy

Exclusion Criteria:

* Stone size < 2 cm
* bilateral ureteral stones
* incomplete stone removal due to impacted stones
* failed ureteroscopic access to the stone
* stone migration to the kidney
* pregnancy
* active urinary tract infection
* solitary kidney
* ureteral stent placed preoperatively
* severe mucosal injury or perforation
* suspected additional ureteral pathology such as ureteral stricture
* urothelial carcinoma or polyp.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score (VAS) | 1 week
  Visual Analog Score (VAS) for flank pain and dysuria score, urgency, frequency, suprapubic pain, hematuria, analgesia requirement, operative time, re-hospitalization, and return to normal physical activity. This is a widely-used scale. It a unidimensional measure of pain intensity. It is administered as a straight horizontal line orientated from the left (worst) to the right (best) , where the patient indicates their situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan